CLINICAL TRIAL: NCT06287216
Title: Preliminary Evaluation of a Mental Health Program: a Comparison Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024001
Record Dates: First submitted 2024-02-05; First posted 2024-03-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-03

CONDITIONS: Mental Wellbeing
MeSH Terms: interventions — Mental Health; Self Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Hygiene Group (Experimental): This is the group participating in the mental hygiene challenge that is willing to give informed consent and conduct pre-post as well as daily well-being surveys.
  Interventions: Behavioral: Mental Hygiene
- Self-Care Group (Active Comparator): Similar to the above, instead of recommending mental hygiene, the investigators will be recommending daily self-care, and offer standard government issued resources, as well as resources from other reputable organizations.
  Interventions: Behavioral: Self-Care

INTERVENTIONS:
Behavioral: Mental Hygiene — Mental hygiene are daily evidence based practices that support mental wellbeing.
  Arms: Mental Hygiene Group
Behavioral: Self-Care — Instructed to do 10 minutes of self-care daily.
  Arms: Self-Care Group

SUMMARY:
The mental hygiene challenge is a Royal Ottawa Health Care Group led initiative to engage the staff, clients and community members to attend to their mental well-being by way of practicing mental hygiene activities for 10 min on a daily basis, throughout the month of March. Participants are encouraged to choose one or many of the practices recommended and do them for about 10 minutes a day. Participants are encouraged to make it their own, in that they can combine the practice or tailor them in a way that suits them best. When signing up for the challenge, participants receive free access to a toolkit with brief outlines and instructional videos on various mental hygiene practices.

Study investigators also encourage participants to divide the 10 minutes in whatever way best works for them, such as 10 minutes all at once, 5 minutes twice, or even 2 minutes five times. This study aims to expand on the work that was done in 2022 and 2023, when the World Health Organization - 5 Wellbeing Index (WHO-5) and the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) were collected from participants to ascertain the impact of mental hygiene, by way of including a control group.

DETAILED DESCRIPTION:
Although mental hygiene is a relatively novel idea, the term can be found in the early 20th century literature. Tremblay et al. {2021) essentially reintroduced the concept and proposed its framework in the scientific literature.

Within public health guidelines, there are standard recommendations given to the public in terms of maintenance of various dimensions of their health. For example, the Canadian Dental Association recommends 2 minutes of teeth brushing twice daily. The World Health Organization (WHO) recommends 150 minutes of moderate physical activity per week for the average adult to support physical health. Showering daily, and frequent hand washing have become embedded in public awareness. As of yet, there is no such well-defined equivalent vis-à-vis mental health in terms of a standardized universal recommendation. Tremblay et al. (2021) proposed a mental hygiene framework that seeks to address this gap and move towards a standardized public facing mental health recommendation equivalent to those that already exist for other dimensions of health. The mental hygiene toolkit is free, accessible and provided through a social equity lens so that anyone from any walk of life can engage in mental wellness without barriers such as cost or availability of time. The preliminary program evaluation findings of the survey data for both years (2022 and 2023) showed a promising signal, which is prompting the investigators to prepare this study that will be built into the 2024 Mental Hygiene Challenge that will involve a control group. It is imperative to continue acquiring empirical data on the impact daily mental hygiene practices has on one's mental wellbeing.

The mental hygiene framework is grounded in 5 main categories of mental training activities. They include: meditation (mindfulness and other techniques), positive psychology interventions, self-directed cognitive behavioral therapy exercises (CBT), pro-social prayer (referring to prayers of thanks and praying for others vs. ritualist/obligatory and supplication prayers), and nature exposure.

The investigators' objective is to gain a better understanding of the impact the mental hygiene challenge has on the wellbeing of its participants for the upcoming Mental Hygiene Challenge of March 2024. In order to do that, the investigators aim to conduct pre-post wellbeing surveys using validated psychometric measures for participants of the challenge. Moreover, the investigators intend to conduct the same pre-post wellbeing survey approach with a control group who will be given standard self-care recommendations. The comparison of the two groups will offer insight on the impact mental hygiene has on those who participate daily.

The investigators overall objective is to determine the impact on mental wellbeing as measured by the WHO-5 and WEMWBS that the mental hygiene challenge of March 2024 will have on its participants. Specifically, the investigators aim to:

* Test the hypothesis that there is a statistically significant change (increase) in the mental wellbeing scores for those that completed the challenge and participated daily.
* To test the hypothesis that the change (increase) in pre-post wellbeing scores in the mental hygiene group will be statistically significantly higher compared to any pre-post change in wellbeing scores of the control group.
* Test the association between participation level and post wellbeing scores. Participation levels will be measured by asking in the post survey how many days they participated in mental hygiene (or self-care) as well as indexing the number of completed daily surveys as an indicator of participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* can speak English

Exclusion Criteria:

* Have previously participated in the mental hygiene challenge (exclusion for the control group).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in level of mental wellbeing as measured by the World Health Organization (WHO)-5 wellbeing index. | Over approximately a 30 day period.
  The psychometric index will be collected before and after the 30 days of mental hygiene or self-care. Higher scores indicate better outcomes (min score =0, max score =25).
Change in level of mental wellbeing as measured by the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Over approximately a 30 day period.
  The psychometric index will be collected before and after the 30 days of mental hygiene or self-care. Higher scores indicate better outcomes (min score = 14, max score = 70).

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No